CLINICAL TRIAL: NCT02974712
Title: The Effects of Two Induction Means on Emergence After General Anesthesia for Elderly Patients Undergoing Transurethral Endoscopic Operation
Brief Title: The Effects of Two Induction Means on Emergence After General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20161114
Record Dates: First submitted 2016-11-14; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Mean Arterial Pressure; Heart Rate
Keywords: Arterial blood gases; MAP; HR
MeSH Terms: interventions — Fentanyl; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): After routine Induction, fentanyl was administrated.
  Interventions: Drug: Fentanyl
- Saline (Placebo Comparator): After routine Induction, same volume saline was administrated.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Fentanyl
  Arms: Fentanyl
Drug: Saline
  Arms: Saline

SUMMARY:
This study aims to investigate the effects of different methods of administration on emergence period after laryngeal mask anesthesia in elderly patients undergoing transurethral endoscopic operation

ELIGIBILITY:
Inclusion Criteria:

* ASA level I or II,
* Aged from 65 to 79,
* With a duration of anesthesia <90 min.

Exclusion Criteria:

* Chronic obstructive pulmonary diseases (COPD),
* Severe heart disease,
* Difficult airway
* Liver and kidney dysfunction,
* Cerebrovascular disease,
* Bleeding volume >20 ml.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) | One hour after surgery

SECONDARY OUTCOMES:
Lengths of stays in the Post anesthesia care unit(PACU) | One hour after surgery